CLINICAL TRIAL: NCT04889898
Title: Home Telemonitoring of Bulbar Function by Acoustic Measurement of Swallowing and Speech Sounds in ALS
Brief Title: Remote Speech and Swallowing Assessment in ALS
Status: Active, not recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Penn State University (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrew Geronimo, Assistant Professor, Neurosurgery, Milton S. Hershey Medical Center
Other Study IDs: STUDY00016872
Record Dates: First submitted 2021-05-07; First posted 2021-05-17 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: telemonitoring; digital health; mobile health; dysphagia; dysarthria
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Deglutition Disorders; Dysarthria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ALS Patients: All ALS patients will be enrolled in this arm, which involves a combination of clinical and home-based assessments of speech and swallowing.
  Interventions: Device: Digital recording of speech and swallow sounds using the Beiwe Digital Health App on a personal smartphone; Radiation: Modified Barium Swallow Study (MBSS); Behavioral: Speech Intelligibility Test (SIT)
- Listeners: Healthy listeners will be recruited to listen to the audio recordings of patients in the study in order to judge the intelligibility of their speech.
  Interventions: Behavioral: SIT Scoring

INTERVENTIONS:
Device: Digital recording of speech and swallow sounds using the Beiwe Digital Health App on a personal smartphone — [Patients only] Weekly completion of audio recordings of speech and swallowing performed at home by the subject using the study smartphone application on their personal device.
  Groups: ALS Patients
Radiation: Modified Barium Swallow Study (MBSS) — [Patients only] MBSS is an instrumented evaluation of oropharyngeal swallowing function that is performed using videofluoroscopy.
  Other Names: Videofluoroscopic Swallowing Study (VFSS)
  Groups: ALS Patients
Behavioral: Speech Intelligibility Test (SIT) — [Patients only] The SIT is a standardized test for measuring speech intelligibility.
  Groups: ALS Patients
Behavioral: SIT Scoring — [Listeners only] Listeners will judge the intelligibility of speech recordings made by patients in the study.
  Groups: Listeners

SUMMARY:
The investigators propose a longitudinal home study of ALS patients to measure the severity of speech and swallowing (bulbar) impairment via a smartphone-based, remote speech and swallow assessment (rSSA). The study is designed to assess the feasibility and validity of such a monitoring intervention. Furthermore, it is proposed that regular monitoring of these two bulbar processes may shed light on their co-evolution over the course of ALS.

DETAILED DESCRIPTION:
Most individuals with ALS experience bulbar function deterioration over the course of the disease which impacts their quality of life significantly. Furthermore, in some patients, bulbar symptoms are an initial presenting symptom of ALS. Identifying these changes, which may be rapid in some individuals, is complicated by the recent acceleration of virtual care delivery.

The investigators propose a longitudinal home study of ALS patients to assess bulbar progression via a smartphone-based, self-administered remote speech and swallow assessment (rSSA). The overall hypothesis is that this monitoring protocol can be used in a way that, 1) is satisfactory to the patient, 2) performs at least as well as standard clinical measures of dysarthria and dysphagia, and 3) resolves the development of emergence of speech and swallowing pathologies in ALS.

ELIGIBILITY:
Inclusion Criteria:

Patients

1. At least 18 years of age
2. Possess a diagnosis of ALS (definite, probable, probable laboratory-supported, or possible by El Escorial criteria [35])
3. Have symptom onset within the last 3 years
4. Demonstrate a score of 2 or 3 in either the speech (item #1) or swallowing (item #3) components of the ALSFRS-R at time of enrollment
5. Demonstrate decline in bulbar function prior to enrollment, measured by a reduction of at least 1 point on either the speech or swallowing components of the ALSFRS-R in the 6 months prior to enrollment. If 6 months of data is not available, an estimate of the change in ALSFRS-R will be calculated from the time of symptom onset.
6. Have a life expectancy ≥ 6 months as determined by the attending neurologist
7. Be fluent in written and spoken English
8. Possess a smartphone capable of running the study application
9. Follow up in the Penn State Hershey multidisciplinary ALS clinic over next 6 months
10. Be able to visit the study site for in-person procedures at weeks 0 and 24

Listeners

1. Between 18 and 40 years of age
2. Native speakers of American English 2.3. Currently residing within the United States. 3.4. Hearing within normal limits, as defined by self report.

Exclusion Criteria:

Patients

1. Possess a co-existing neurological or psychiatric illness that, in the opinion of the study team, exclude the subject from participation
2. Demonstrate clinically significant dementia, as determined by the ALS study neurologist
3. Possess abnormal speech or swallowing processes due to a condition independent of their ALS diagnosis

Listeners

1. Have an identified speech, language, learning, or neurological disorders per self-report
2. Experience communicating with people with motor speech disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population 1: Patients with ALS Population 2: Healthy Listeners
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Digital recording of speech and swallow | weekly for 24 weeks
  Audio recordings of speech tasks and spontaneous swallowing task

SECONDARY OUTCOMES:
MBS Impairment Profile (MBSImp) | Weeks 0 and 24
  Standardized scoring for the MBSS in 17 domains. Domains are aggregated in to scores for Oral Impairment (0-22), Pharyngeal Impairment (0-29), and Esophageal Impairment (0-4), with higher scores indicating impaired function.
Speech Intelligibility Task (SIT) Intelligibility listener scoring | Weeks 0, 12, and 24
  Listeners will score the intelligibility of patient SIT recordings
ALS Functional Rating Scale - Revised (ALSFRS-R) | Weeks 0, 12, and 24
  ALS Specific Assessment of physical function ranging from 0-48, with 48 being normal function.
Center for Neurological Study - Bulbar Function Scale (CNS-BFS) | Weeks 0, 4, 8, 12, 16, 20, and 24
  Self-administered rating scale for speech (7-49) and salivation (7-35) functions, with high scores indicating impaired function.
Mann Assessment of Swallowing Ability (MASA) | Weeks 0, 12, and 24
  A standard clinical swallowing assessment performed by the speech-language pathologist. Scores range from 38-200, with lower scores indicating higher impairment.
EAT-10 Questionnaire | Weeks 0, 12, and 24
  A self-reported assessment of eating and swallowing function. Scores range from 0-40, with higher scores indicating higher impairment.
Forced Vital Capacity (FVC) | Weeks 0, 12, and 24
  A standard clinical respiratory assessment of vital capacity
Maximal Inspiratory Pressure (MIP) | Weeks 0, 12, and 24
  A standard clinical respiratory assessment of inspiratory strength

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Geronimo, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Hershey Medical Center ALS Clinic, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No